CLINICAL TRIAL: NCT02159391
Title: The Efficacy of Brief Motivational Interviewing for Trauma Patients Related to Alcohol or Other Abuse Drugs.
Acronym: MOTIVA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundación Pública Andaluza para la Investigación Biomédica Andalucía Oriental (Other)
Collaborators: Universidad de Granada (Other); Andaluz Health Service (Other Government)
Responsible Party: Principal Investigator, Raquel Vilar Lopez, Prof. Experimental Psychology Department, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI 0691-2013; PI-0691-2013 (Other: JUNTA DE ANDALUCIA)
Record Dates: First submitted 2014-06-06; First posted 2014-06-09 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: AODD and AODR Disorder
Keywords: Accident Prevention; Alcohol Drinking; Substance-Related Disorders; Motivational Interviewing; Adult; Humans; Intervention Studies; Recurrence; Risk Factors; Trauma Centers; Wounds and Injuries/epidemiology; Wounds and Injuries/etiology*; Wounds and Injuries/prevention & control*
MeSH Terms: conditions — Alcohol Drinking; Substance-Related Disorders; Recurrence; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Intervention (No Intervention): A standard intervention will be performed by nursing staff during hospital admission. Written information about the consequences of driving under the influence of alcohol and/or drugs will be provided. No psychological intervention.
- Brief Motivational Interview (Experimental): A Brief Motivational Interviewing will be performed during hospital admission by a psychologist experienced with this intervention.
  Interventions: Behavioral: Brief Motivational Interview

INTERVENTIONS:
Behavioral: Brief Motivational Interview — The Brief Motivational Interview implies an empathic interviewing style which (i) recognizes, examines and tries to resolve the patient´s ambivalence to facilitate behavioral change, (ii) promotes self-efficacy, (iii) allows flexibility in strategies, including short-term aims to reduce consumption and decrease damage linked to this consumption (like road accidents), (iv) works to reduce the patient's resistances, and (v) provides individualized feedback, if deemed appropriate, to promote recognition of the problem and cognitive restructuring.
  Arms: Brief Motivational Interview

SUMMARY:
The purpose of this study is to determine whether the Brief Motivational Interview will produce a significantly reduction in risk behavior than usual treatment 3 months after discharge from hospital in people who have survived a traumatism.

DETAILED DESCRIPTION:
Objectives:

1. To determine the efficacy of Brief Motivational Interview against an usual hospital treatment (no psychological treatment) in patients who have suffered an accident under the influence of drugs (1) to reduce risk behaviors and drug consumption and (2) to increase motivation to change behavior and risk perception.
2. To investigate the mediating role of impulsive personality and decision making in the impact of Brief Motivational Interview on reduction of risk driving.
3. To assess the economic viability of the results of Brief Motivational Interview through a cost-utility analysis.

ELIGIBILITY:
Inclusion Criteria:

* Trauma patients who have had: 1) A road crash, 2) A sport injury, 3) Occupational accident.
* Tested positive on alcohol and/or other abuse drugs tests.

Exclusion Criteria:

* Cognitive or brain-damage that prevent assessment and Brief Motivational Interview
* Psychopathological disorders
* Residence status that prevents follow-up (residence outside of Spain, homeless).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-03 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Risk behavior | Baseline, month 3.
  Measure with Short Driver Behaviour Questionnaire (SDBQ) and Domain-Specific Risk-Taking (DOSPERT)

SECONDARY OUTCOMES:
Alcohol and Other Drug consumption | Baseline, month 3.
  Measure with Timeline Followback (TLFB), Interview for Research on Addictive Behavior (IRAB) and Audit Test.
Motivation to change | Baseline, post-intervention, month 3
  Measure with SOCRATES-8
Risk perception | Baseline, post-intervention, month 3.
  Risk perception questionnaire, perceived risk of alcohol and drug (EDADES).
General Health | Baseline, month 3.
  Measure with SF6D

OTHER OUTCOMES:
Risk Taking and Impulsive Behavior | Baseline, month 3.
  Measure with Impulsive Behavior Scale (UPPS-P) and Self-efficacy questionnaire
Real-life decision making | Baseline, month 3.
  Iowa Gambling Task (IGT)

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Vilar, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Hospital Virgen de las Nieves, Granada, Andalusia, Spain